CLINICAL TRIAL: NCT05903703
Title: Clinical Study of Capeline Combined With Gemcitabine in the Treatment of Pancreatic Cancer
Brief Title: Canagliflozin With Gemcitabine in Pancreatic Carcinoma
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhang Xiaofeng,MD (Other)
Collaborators: College of Pharmaceutical Sciences at Zhejiang University (Unknown); The Innovation Institute for Artificial Intelligence in Medicine, Zhejiang University (Unknown)
Responsible Party: Sponsor-Investigator, Zhang Xiaofeng,MD, chief physician, First People's Hospital of Hangzhou
Organization: First People's Hospital of Hangzhou (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20230519
Record Dates: First submitted 2023-05-19; First posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Canagliflozin; Gemcitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Canagliflozin and Gemcitabine (Experimental)
  Interventions: Drug: Canagliflozin and Gemcitabine
- standard cisplatin (Active Comparator)
  Interventions: Drug: Gemcitabine

INTERVENTIONS:
Drug: Canagliflozin and Gemcitabine — on the first, 8th and 15th day of treatment, patients were given intravenous drip of 1000mg/m2 gemcitabine, and 21 days was a course of treatment, lasting for 6 courses.
  Take 400mg canagliflozin orally every day, and continue to use it until the end of chemotherapy. According to the patient's tolerance to disulfiram, the dose of canagliflozin can be re-evaluated during the treatment, and the highest dose is 125mg per day. The clinical symptoms, signs and adverse reactions of patients were observed, and the treatment effect of patients was evaluated after two consecutive cycles with 4 weeks as a cycle
  Arms: Canagliflozin and Gemcitabine
Drug: Gemcitabine — on the first, 8th and 15th day of treatment, patients were given 1000mg/m2 gemcitabine intravenously, and 21 days was a course of treatment, lasting for 6 courses.
  Arms: standard cisplatin

SUMMARY:
Gemcitabine-based chemotherapy or combination with FOLFIRINOX is the leading treatment of pancreatic cancer. However, the overall response rate of pancreatic cancer to gemcitabine is less than 20%. Resistance to gemcitabine is the most important reason. There is an urgent need to develop new combination therapies to improve the efficiency of chemotherapy, avoid toxicity limitations, and improve the overall prognosis of pancreatic cancer. At present, it has been found that canagliflozin can reduce the expression level of PD-L1 in pancreatic cancer and restore the vitality of CD8+ T cells. Canagliflozin combined with gemcitabine may improve the efficiency of chemotherapy.

ELIGIBILITY:
1. Inclusion criteria: # Age ≥18 years old; #Metastatic or unresectable pancreatic cancer is confirmed through histology or cytology; # Estimated survival time > 3 months; # Without any chemotherapy treatment or more than one month from the end of the last chemotherapy course; #ECOG physical status score 0-2;
2. Exclusion criteria: # patients who had allergic reaction to therapeutic drugs; # patients with other types of cancer; # Patients with severe diseases of heart, liver, kidney, etc.; (4) gastrointestinal dysfunction or unable to oral medication.
3. Shedding/eliminating criteria: exiting in the midway; Lost to follow-up during the follow-up period; Treatment was not continued according to the treatment protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation the clinical complete response (CR) at 6 weeks intervals | 18 weeks
  The tumor lesion in our patient completely resolved and lasted for ≥4 weeks, and no new lesion appeared
Evaluation the clinical partial response (PR) at 6 weeks intervals | 18 weeks
  the overall reduction in the longest diameter of the tumor focus is > 50% and it can be maintained for at least 4 weeks, with no new focus emerging
Evaluation the clinical stable disease (SD) at 6 weeks intervals | 18 weeks
  the overall reduction or increase of the longest diameter of the tumor lesion is < 50% or < 25%, and the duration is > 4 weeks; no new lesion appears
Evaluation the clinical disease progression (PD) at 6 weeks intervals | 18 weeks
  the combined increase in the longest diameter of the tumor lesion is ≥25%, or a new lesion appears

CONTACTS AND LOCATIONS:
Locations (1):
- Hangzhou first people's Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No